CLINICAL TRIAL: NCT00239174
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose, Multi-Center Study Evaluating the Efficacy and Safety of Four Doses of SR147778 in Obese Patients
Brief Title: A Multicenter Study to Evaluate the Efficacy and Safety of of Four Doses of SR147778 in Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI5029
Record Dates: First submitted 2005-10-13; First posted 2005-10-14 (Estimated); Last update posted 2008-12-10 (Estimated); Status verified 2008-12

CONDITIONS: Obesity
Keywords: obesity
MeSH Terms: conditions — Obesity | interventions — surinabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR147778

SUMMARY:
The purpose of this study is to assess the effect of SR147778 on weight loss over a period of 24 weeks when prescribed with a hypocaloric diet in obese patients. The secondary objective is to assess the safety and tolerability of SR147778 and to assess the effect of SR147778 on several secondary parameters (such as waist, metabolic parameters) over a period of 24 weeks when prescribed with a hypocaloric diet in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must voluntarily sign the informed consent,
* Patients must be male or female and aged 18 to 65 years,
* Patients must be able to follow verbal and written instructions,
* Female patients of childbearing potential (pre-menopausal women) must have a confirmed negative urine b-hCG pregnancy test prior to enrollment and Baseline Visit. They must use an acceptable double method of birth control (e.g., oral or implanted contraceptive therapy, or IUDs, plus a barrier such as condom, diaphragm or spermicide) throughout the study, and accept to repeat urine b-hCG pregnancy test at designated visits,
* Patients must have a BMI >=30 and <= 40 at screening
* Patients must have had a stable weight (variation of less than 5 kg during the 90 days preceding the Screening Visit)
* Patients must have shown to be compliant to dietary recommendations between the Screening and the Baseline Visits
* Patients' physical examination, laboratory evaluations, 12-lead ECG must be within normal limits (with the exception of abnormalities considered as clinically insignificant in the opinion of the Investigator and the Center Monitor), or within predefined limits for hemoglobin (>= 11 g/dL), total cholesterolemia (<= 3 g/L, i.e. 7.7 mmol/L), triglyceridemia (<= 7 g/L, i.e. 7.9 mmol/L), fasting glycemia (<= 1.6 g/L, i.e. 8.9 mmol/L), and hemoglobin A1c (<= 8%).

Exclusion Criteria:

* Female patients who are pregnant or lactating,
* Patients who are considered by the Investigator to be unsuitable candidates for receipt of an investigational drug,
* Myocardial infarction within 12 months,
* Hypertension (SBP > 160 mmHg; DBP > 95 mmHg),
* Secondary hypertension- Confirmed heart rate < 60 beats/minute,
* Type 1 diabetes, or treated with insulin
* History or presence of pancreatitis,
* History or presence of clinically significant cardiac valve disorder or abnormal cardiac echography.
* History or concurrent DSM-IV bulimia or anorexia nervosa,
* Patients with mental retardation or any clinically significant psychiatric disorder (including organic mental disorder) other than mild mood or anxiety,
* History (during the past six months) or concurrent DSM-IV substance abuse or dependence (excluding nicotine and caffeine as far as patient agrees not to modify her/his consumption throughout the study),
* Severe or multiple drug allergies,
* Any disorder that may interfere with drug absorption, metabolism distribution or excretion,
* Presence of any clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, endocrine, dermatological or respiratory disease, or any other medical condition that might interfere with the evaluation of study medication,
* Prolonged QTcB: > 450 msec for men and > 470 msec for women.
* Patients who test positive for any illicit drug included in the urine drug screen (THC) at the Screening or the Baseline Visit. Patients positive for benzodiazepines only may be admitted, if prescribed with stable dose regimen.
* Patients who test positive at the Screening Visit for hepatitis B surface antigen, hepatitis C antibody, or ALT and/or AST > 2 x upper limit of normal,
* Hb < 11g/dL, fasting glycemia > 1.6 g/L i.e. 8.9 mmol/L, HbA1c > 8%, total cholesterolemia > 3 g/L i.e. 7.7 mmol/L, or TG > 7 g/L i.e. 7.9 mmol/L, creatinemia > 150 mmol/l- Patients who have received anti-obesity drugs or other drug(s) or preparation(s) including herbal for weight reduction within three months of Screening Visit,
* Thyroid therapy, except on replacement therapy.
* Patients using nicotine substitutes or taking bupropion,
* Treated with antidepressant or neuroleptics drug(s) for more than one week within three months of Screening Visit,
* Treated with non selective systemic antihistamines
* Systemic corticosteroids or inhaled corticosteroids
* Treated with potent inhibitors of CYP3A4
* Consuming more than 20 g/day of alcohol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2004-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Weight loss at 6 months.

SECONDARY OUTCOMES:
Waist circumference,lipid parameters,glycemic parameters,metabolic syndrome,blood pressure,adipokines,CRP,IL-6,IL-2,patient satisfaction,food behavior,daily caloric intake, and dietary compliance at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Laville, MD, Principal Investigator — Hôpital Edouard Herriot, Endocrinologie-Diabète-Nutrition, 5 Place d'Arsonval, 69437 LYON cedex 03, France
Locations (5):
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Barcelona, Spain

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com